CLINICAL TRIAL: NCT05316402
Title: Sun Exposure for Outdoor Athletes in Mayotte and Reunion Island
Acronym: EXSPOSOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021/CHU/39
Record Dates: First submitted 2022-03-14; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-02

CONDITIONS: Sun Exposure
Keywords: Sun Exposure, sportsmen
MeSH Terms: interventions — Radiometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- training on the risks associated with sun exposure (Experimental): power point on the risks associated with sun exposure
  Interventions: Other: training on the risks associated with sun exposure; Other: dosimetry

INTERVENTIONS:
Other: training on the risks associated with sun exposure — 15-minute power point and presentation on the risks of sun exposure
Other: dosimetry — dosimetry

SUMMARY:
The UV index in Mayotte and Reunion is greater than 14, eight months out of 12. This index decreases linearly over the period from mid-April to mid-August where it can drop to reach an index of 8 in the month of July. The inhabitants are therefore exposed to a maximum intensity of UV radiation according to the WHO.

The World Health Organization (WHO) recommends extreme precautions for indices greater than 11 (avoid exposure between 11 a.m. and 3 p.m. (GMT+3 hours), stay in the shade, wear a t-shirt, sunglasses, hat and sunscreen).

Sun exposure is a major risk factor in the development of skin cancer, basal cell cancer, squamous cell cancer and cutaneous melanoma. It is also the cause of premature aging of the skin. Moreover, it causes ocular complications such as the occurrence of cataracts and this without distinction of skin phenotype.

There is currently no prevention campaign on the risks of sun exposure in Mayotte or Reunion for adults, while many risky behaviors are observed both in the professional field and during leisure activities. In order to better understand risk-taking and choose appropriate awareness-raising tools, it is necessary to identify the knowledge, attitudes and practices (KAP) of these populations in terms of risk of sun exposure and to measure the impact of solar prevention education actions.

ELIGIBILITY:
Inclusion Criteria:

* Live in Mayotte or Reunion island
* 18 years old,
* Practice outdoor sports > 4 hours per week in one of the identified sports associations
* Belong to the list of targeted associations

Exclusion Criteria:

* Person deprived of liberty by judicial or administrative decision, minor, and person subject to a legal protection measure: guardianship or curators
* Person not wishing to participate
* No one speaking any of the following languages: English / French / Shimaore / Kibushi / Creole or Comorian
* Person who cannot be followed during the 6 months of the study
* Inability to answer the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Improve the knowledge of photo-exposed sportsmen on the risks associated with exposure to the sun | 6 month
  knowledge quiz

SECONDARY OUTCOMES:
Assess the change in attitudes and practices of photo-exposed sportsmen | 6 month
  attitudes and practices of photo-exposed workers quiz
fitzpatrick scale : classification of skin types (phototype I to VI) | 6 month
  association between phototype and knowledge level
knowledge questionnaire on the risks of sun exposure | 6 month
  association between phototype and knowledge level
Obtain UV dosimetry data by occupation to confirm risk exposure during working hours. | 6 month
  dosimetry data

CONTACTS AND LOCATIONS:
Locations (2):
- Mayotte, Chirongui, Mayotte
- Reunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No